CLINICAL TRIAL: NCT04601922
Title: Qualitative Study of Potential Barriers and Solutions to Long Term Cardiovascular Risk Prediction in the Emergency Department
Brief Title: Qualitative Study of Long Term Cardiovascular Risk Prediction in the Emergency Department
Status: Completed | Type: Observational
Sponsor: University of Manchester (Other)
Collaborators: Royal College of Emergency Medicine (Other)
Responsible Party: Principal Investigator, Richard Body, Professor of Emergency Medicine, University of Manchester
Other Study IDs: NHS 001549
Record Dates: First submitted 2020-10-09; First posted 2020-10-26 (Actual); Last update posted 2022-07-05 (Actual); Status verified 2022-06

CONDITIONS: Cardiovascular Diseases; Cardiovascular Risk Factor; Emergencies
MeSH Terms: conditions — Cardiovascular Diseases; Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Emergency Medicine Consultants
  Interventions: Other: Semi-structured interview
- General Practitioners
  Interventions: Other: Semi-structured interview
- Acute care nursing staff
  Interventions: Other: Semi-structured interview
- Patients presenting with suspected cardiac chest pain
  Interventions: Other: Semi-structured interview

INTERVENTIONS:
Other: Semi-structured interview — The interview will have the audio recorded, and will explore the ideas of each participant around long term cardiovascular care pathways

SUMMARY:
One of the most common presentations to ED is chest pain, with the rapid rule out of heart attacks in the emergency department being common place. This moves a new onus of responsibility to the ED; the care of long term heart disease. A study conducted locally demonstrated that patient's with a heart attack ruled out felt the 'what next' question is not answered sufficiently at present. The strength of this opportunity is re-enforced by studies suggesting that chest pain presents a teachable moment where patients are more accepting of advice.

The study's overarching goal is to improve heart disease care (cardiovascular disease).The early warning signs for heart disease can be detected and treated enabling patients to live longer and healthier lives.

This is where it is believed that the Emergency Department (ED) can improve, EDs already collect the vast majority of data required to detect these early warning signs. In the United Kingdom more than 23.8 million attendances were registered last year, and ED is currently underusing a large amount of patient data of potentially great value to the population.

The study aims to explore the best way to use this long term heart disease prediction; how to communicate it to patients, who prescribes the necessary medication, who issues lifestyle advice, and who follows it up.

The investigators intend to answer these questions with a series of semi-structured interviews. The study will comprise of initial semistructured interviews made up of emergency medicine consultants, general practitioners, nurses, and patients. Then building on the knowledge gained from the initial interviews it is planned to build a prototype care pathway that will be explored in the second set of interviews.

Funded by The Royal College of Emergency Medicine

Ethical approval by the UK's HRA REC - 19/WA/0312

ELIGIBILITY:
Inclusion Criteria:

* Genaral Practitioner / Emergency medicine consultant consultant /acute care nurse OR
* emergency department patients with low risk chest pain.

These patients are deemed low risk by a predictive algorithm that was validated in more than 10,000 and has subsequently been used in clinical practice safely in over 7,000 patients. Once deemed low risk they are then transferred to an ambulatory care unit where they receive further assessment.

Exclusion Criteria:

* The participants can not attend at least one of the semi-structured interviews
* Not fluent in English language
* The ambulatory ward patient's clinical condition has deteriorated or is severe to the extent that participating in the research would (a) interfere in their clinical care, or (b) that participating would be too strenuous. This will be judged by the nursing staff on the ambulatory care unit, and the clinical academics interviewing the patients.
* Unwilling to take part

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: * Genaral Practitioner
  * Emergency medicine consultant consultant
  * acute care nurse
  * emergency department patients with low risk chest pain.
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2020-09-15 (Actual); Primary Completion 2022-01-18 (Actual); Study Completion 2022-01-18 (Actual)

PRIMARY OUTCOMES:
Experience and views of barriers and solutions to the provision of preventative medicine in the emergency department. | 30-45 minutes
  Through semi-structured interviews the study will focus specifically on the prevention of cardiovascular disease in those patients presenting with chest pain. Qualitative software will be used to thematically analyse the interviews.
Prototype care pathways for prevention of long term cardiovascular disease | through study completion, an average of 1 year
  The study is seeking through co-design to develop prototype care pathways for the prevention of cardiovascular disease.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Body, MbChB, PhD, FRCEM, Study Director — University of Manchester
Locations (1):
- Manchester Royal Infirmary, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Ethical approval register — https://www.hra.nhs.uk/planning-and-improving-research/application-summaries/research-summaries/a-qualitative-study-of-long-term-cardiovascular-risk-prediction-in-ed/